CLINICAL TRIAL: NCT05668000
Title: Self-Monitoring Using Mobile App for Reduction of Rehospitalization and Mortality in Heart Failure (SMART-HF)
Brief Title: Mobile App for Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: KT Corporation (Industry)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART-HF
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIDA/KT-app with devices (Experimental): AIDA/KT-app with devices : with device link and with feedback
  Interventions: Other: Bluetooth-connected monitoring devices and a feedback system; Other: Mobile application
- AIDA/KT-app only (Placebo Comparator): AIDA/KT-app only : no device link or no feedback
  Interventions: Other: Mobile application

INTERVENTIONS:
Other: Bluetooth-connected monitoring devices and a feedback system — AIDA/KT-app with devices and feedback:
  The mobile application provide self-management interventions with devices including sphygomanometer and body water meter and a feedback system
  Arms: AIDA/KT-app with devices
Other: Mobile application — The mobile application provide only self-management interventions.

SUMMARY:
The investigators developed a mobile health platform to self-management in HF. The aim of this study is to evaluate whether this smartphone app-based intervention can improve symptoms of HF when compared to usual care in HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older hospitalized for acute heart failure.
* Patients who have obvious symptoms or sign of HF at admission
* N-terminal prohormone of brain natriuretic peptide (NT-proBNP) ≥400 pg/mL or brain natriuretic peptide (BNP) ≥100 pg/mL.
* participants should be able to use smartphone well.

Exclusion Criteria:

* Patients who have baseline systolic blood pressure <90 mmHg or resting heart rate <50 beats per minutes
* Patients who cannot use smartphone
* Patients who had cardiac implantable electronic device will be excluded

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
HF symptom by application scores. | 4 weeks
  the mean value of scores of dyspnea, fatigue, and ankle edema stored in app by participants will be evaluated.
  Range 0(no symptom) - 3(severe symptom)
HF symptom by questionnaire | 4 weeks
  The degree of dyspnea will be evaluated by questionnaire. Range: 0(worst)-10(best)

SECONDARY OUTCOMES:
Composite outcome | 4 weeks
  including death, rehospitalization, and unscheduled HF visit
Application satisfaction score | 4 weeks
  The satisfaction score will be evaluated by questionnaire. Range: 0(worst)-10(best)
change in body water composition f | 4 weeks
  the change in body water composition from baseline to the last measurement in the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, Study Chair — Seoul National Univeristy Bundang Hospital
Locations (7):
- South Korea (7):
  - Keimyung University Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam
  - Catholic University college of medicine, Seoul
  - Korea Univ. Guro hospital, Seoul
  - Samsung medical center, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Wonju Severance Hospital, Wŏnju

REFERENCES:
- [Derived] Yoon M, Lee S, Choi JY, Jung MH, Youn JC, Shim CY, Choi JO, Kim EJ, Kim H, Yoo BS, Son YJ, Choi DJ. Effectiveness of a Smartphone App-Based Intervention With Bluetooth-Connected Monitoring Devices and a Feedback System in Heart Failure (SMART-HF Trial): Randomized Controlled Trial. J Med Internet Res. 2024 Apr 29;26:e52075. doi: 10.2196/52075. PMID 38683665